CLINICAL TRIAL: NCT00430820
Title: Discovery of New Circulating Biomarkers of Coronary Atherosclerosis Using Differential Proteomics: the BIOmarkers of CORonary Events (BIOCORE) Study
Brief Title: Discovery of New Circulating Biomarkers of Coronary Atherosclerosis
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Fédération Française de Cardiologie (Other); Société Française de Cardiologie (Other)
Responsible Party: Yannick Vacher, Department Clinical Research of Developppement
Other Study IDs: P060201
Record Dates: First submitted 2007-02-01; First posted 2007-02-02 (Estimated); Last update posted 2010-12-03 (Estimated); Status verified 2009-04

CONDITIONS: Coronary Artery Disease; Acute Coronary Syndromes; Myocardial Infarction; Atherosclerosis
Keywords: Biomarkers; Proteomics; Mass spectrometry; Atherosclerosis; Acute coronary syndromes; Myocardial infarction; Coronary artery disease
MeSH Terms: conditions — Coronary Artery Disease; Acute Coronary Syndrome; Myocardial Infarction; Atherosclerosis

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — biomarqueurs
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: 30 patients
  Interventions: Procedure: per intervention
- 2: 30 patients
  Interventions: Procedure: per intervention
- 3: 30 patients
  Interventions: Procedure: per intervention

INTERVENTIONS:
Procedure: per intervention — per intervention

SUMMARY:
The study hypothesis is that differential proteomic techniques can be used to discover new circulating biomarkers of coronary atherosclerosis in the blood of patients suffering from coronary artery disease (either stable or unstable) who will be compared to a group of patients without coronary artery disease

DETAILED DESCRIPTION:
Hypothesis: Our hypothesis is that coronary atherosclerosis induces both quantitative and qualitative modifications of circulating proteins, which can be captured by a differential proteomic approach applied to serum or plasma samples. Identification of such modifications in the circulating blood of patients with coronary artery disease (versus patients without coronary artery disease) and/or of patients with acute coronary syndromes (versus stable coronary artery disease) may lead to discovery of new biomarkers of coronary atherosclerosis and of atherosclerotic plaque vulnerability.

Objectives:

Primary objective: Identification of new circulating biomarkers of stable and unstable coronary artery disease using a new approach of differential proteomics.

Secondary objectives:

* Evaluation of the diagnostic value of these new biomarkers for the diagnosis of stable and unstable coronary artery disease.
* Comparison of the diagnostic value of these new biomarkers to the diagnostic value of 1) other validated biomarkers of atherosclerosis (eg, CRP, IL-6, CD40L, markers of leukocyte activation, …); and 2) of non-invasive measures of arterial function (eg, carotid artery intima-media thickness, pulse wave velocity, ankle/brachial index, …)
* Description of the relationship between these new biomarkers and major adverse coronary events (death, myocardial infarction, revascularization) during a 12-month follow-up.

Methods:

Uniq center, prospective study. Three groups of patients will be studied. Group 1: Non-ST-elevation acute myocardial infarction; Group 2: Stable coronary artery disease; Group 3: normal coronary arteries and absence of other detectable atherosclerotic lesions.

A new proteomic approach will be applied to serum and plasma samples obtained 1 month after the index hospitalisation. This approach includes 3 steps: 1) equalisation of circulating proteins (expose low-concentration proteins belonging to the "deep-proteome"); 2) Retention chromatography; and 3) protein separation using 2D-electrophoresis and Surface-Enhanced Laser Desorption/Ionisation Time-of-Flight (SELDI-TOF).

Biomarkers with the highest diagnostic value will be subsequently identified using Matrix-Assisted Laser Desorbtion/Ionisation Time-of-Flight (MALDI-TOF) and tandem mass spectrometry (MS/MS).

Perspectives:

Validation of the diagnostic and prognostic values of the new biomarkers discovered and identified using the proteomic approach described above will require development of more straightforward measurement techniques (eg, ELISA), which will be used prospectively or retrospectively in other cohorts of patients with coronary artery disease. Basic studies will be performed in parallel, so as to better understand the role of these new biomarkers in the pathophysiology of atherosclerosis.

ELIGIBILITY:
Inclusion Criteria:

* Group 1 (Non-ST-elevation acute myocardial infarction) :

  * Chest pain less than 48 hours before admission,
  * And modifications of ST-T (no persistent ST elevation) on 12-lead EKG,
  * And elevation of troponin-I >1xN,
  * And presence of ≥1 de novo stenosis(es) >50% located on ≥1 native coronary artery(ies) and successfully treated using percutaneous coronary intervention and stenting.
* Group 2 (Stable coronary artery disease) :

  * Documented myocardial ischemia (stable angina or positive stress test)
  * And presence of ≥1 de novo stenosis(es) >50% located on ≥1 native coronary artery(ies) and successfully treated using percutaneous coronary intervention and stenting.
* Group 3 (Normal coronary arteries) :

  * No history of coronary artery disease, neurovascular disease or peripheral artery disease,
  * And normal coronary angiography performed because of suspected coronary artery disease
  * And absence of significant functional or anatomic abnormalities suggestive of atherosclerosis on non-invasive arterial studies (measurements of intima-media thickness, pulse wave velocity, ankle-brachial index, …).

Exclusion Criteria:

* Group 1 :

  * Preexisting EKG abnormalities (including left bundle branch block) precluding accurate assessment of ST-T changes
* Group 2 :

  * History of acute coronary syndrome
* Groups 1 and 2:

  * Culprit coronary artery stenosis is a restenosis or a stent thrombosis or is located in a bypass graft.
* All groups :

  * Heart failure (NYHA class ≥II)
  * Left ventricular ejection fraction <50%
  * Severe valvular heart disease requiring surgical or percutaneous therapy
  * History of autoimmune, inflammatory or neoplasia diseases ; or infectious disease in the month before admission
  * Life expectancy < 1 year
  * Age <18 years or >80 years
  * Current pregnancy or breast-feeding
  * Homeless or travelers who may not be followed-up
  * Refusal to sign the informed consent form

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Identification de nouveaux marqueurs circulants de l'athérosclérose coronarienne et de ses complications par une nouvelle technique de protéomique différentielle.
  Identification of new parqueurs circulated in coronary artheriosclerosis and complications of the new differentiel technicology
Sampling Method: Probability Sample
Enrollment: 124 (Actual)
Dates: Start 2007-03; Primary Completion 2009-07 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laurent FELDMAN, MD,PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Department of Cardiology, Hopital Bichat, APHP, Paris, France

REFERENCES:
- [Result] Duran MC, Mas S, Martin-Ventura JL, Meilhac O, Michel JB, Gallego-Delgado J, Lazaro A, Tunon J, Egido J, Vivanco F. Proteomic analysis of human vessels: application to atherosclerotic plaques. Proteomics. 2003 Jun;3(6):973-8. doi: 10.1002/pmic.200300389. PMID 12833522
- [Result] Martin-Ventura JL, Duran MC, Blanco-Colio LM, Meilhac O, Leclercq A, Michel JB, Jensen ON, Hernandez-Merida S, Tunon J, Vivanco F, Egido J. Identification by a differential proteomic approach of heat shock protein 27 as a potential marker of atherosclerosis. Circulation. 2004 Oct 12;110(15):2216-9. doi: 10.1161/01.CIR.0000136814.87170.B1. Epub 2004 Jul 12. PMID 15249501
- [Result] Vivanco F, Martin-Ventura JL, Duran MC, Barderas MG, Blanco-Colio L, Darde VM, Mas S, Meilhac O, Michel JB, Tunon J, Egido J. Quest for novel cardiovascular biomarkers by proteomic analysis. J Proteome Res. 2005 Jul-Aug;4(4):1181-91. doi: 10.1021/pr0500197. PMID 16083268
- [Result] Blanco-Colio LM, Martin-Ventura JL, Vivanco F, Michel JB, Meilhac O, Egido J. Biology of atherosclerotic plaques: what we are learning from proteomic analysis. Cardiovasc Res. 2006 Oct 1;72(1):18-29. doi: 10.1016/j.cardiores.2006.05.017. Epub 2006 May 24. PMID 16814757
- [Derived] Ramos-Mozo P, Madrigal-Matute J, Vega de Ceniga M, Blanco-Colio LM, Meilhac O, Feldman L, Michel JB, Clancy P, Golledge J, Norman PE, Egido J, Martin-Ventura JL. Increased plasma levels of NGAL, a marker of neutrophil activation, in patients with abdominal aortic aneurysm. Atherosclerosis. 2012 Feb;220(2):552-6. doi: 10.1016/j.atherosclerosis.2011.11.023. Epub 2011 Nov 25. PMID 22169111